CLINICAL TRIAL: NCT05992675
Title: Air Optix® Night and Day® Aqua Continuous Wear
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: CLD265-N003
Record Dates: First submitted 2023-08-08; First posted 2023-08-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Refractive Errors
Keywords: Contact Lenses; Overnight wear
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- AONDA contact lenses: Lotrafilcon A contact lenses worn in a 30-day, continuous wear modality (lenses worn continuously including overnight) over a period of approximately 3 years
  Interventions: Device: Lotrafilcon A contact lenses
- PV2 contact lenses: Balafilcon A contact lenses worn in a 30-day, continuous wear modality (lenses worn continuously including overnight) over a period of approximately 3 years
  Interventions: Device: Balafilcon A contact lenses

INTERVENTIONS:
Device: Lotrafilcon A contact lenses — CE-marked silicone hydrogel contact lenses
  Other Names: Air Optix® Night and Day® Aqua; AONDA
  Groups: AONDA contact lenses
Device: Balafilcon A contact lenses — CE-marked silicone hydrogel contact lenses
  Other Names: PureVision® 2; PV2
  Groups: PV2 contact lenses

SUMMARY:
The purpose of this retrospective, Post-Market Clinical Follow-Up (PMCF) study is to assess the long term performance and safety of Air Optix® Night and Day® Aqua (AONDA) contact lenses in a real-world setting when worn as 30 days of continuous wear for vision correction.

DETAILED DESCRIPTION:
This is a non-interventional/observational study designed as a retrospective chart review. Study sites will identify charts within their existing databases in a fair and consistent manner. Subjects/charts meeting the eligibility criteria will be enrolled in the study.

The study is designed with one period. The duration of the period includes the Baseline Visit and the Year 3 Visit as follows:

* The Baseline Visit is defined as the first office visit where an eye care professional provided an in-person office biomicroscopy exam to the subject, before or during which a contact lens prescription for AONDA or PureVision 2 (PV2) was released.
* The Year 3 Visit is defined as a visit which occurred 3 years (-2/+8 months) since Baseline during which period the subject was wearing AONDA contact lenses or PV2 contact lenses and a contact lens examination was performed.

The data collection period is defined as any approximately 3-year timeframe since and including 2009.

ELIGIBILITY:
Key Inclusion Criteria:

* Manifest refraction cylinder less than or equal to 0.75 diopter in each eye at baseline
* Best corrected visual acuity of 20/25 or better in each eye at baseline
* At the time of Year 3 Visit, subject was prescribed and wearing AONDA or PV2 contact lenses in both eyes in a 30-day continuous wear modality for at least approximately 3 years
* Baseline Visit and Year 3 Visit charts available

Key Exclusion Criteria:

* Any recurrent history or active anterior segment infection, inflammation, abnormality, or disease contraindicating regular contact lens wear present at baseline
* The use of systemic or ocular medications contraindicating regular contact lens wear at baseline
* History of refractive surgery or irregular cornea
* Slit lamp findings, including signs of pathological dry eye, that would contraindicate regular contact lens wear at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators will enroll charts following a pre-identified process.
Sampling Method: Non-Probability Sample
Enrollment: 1256 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
Distance visual acuity | Year 3
  The subject's chart will be reviewed for distance visual acuity.
Incidence of corneal infiltrative events | Up to Year 3
  The subject's chart will be reviewed for incidences of corneal infiltrative events occurring after the Baseline Visit exam.
Incidence of microbial keratitis | Up to Year 3
  The subject's chart will be reviewed for incidences of microbial keratitis occurring after the Baseline Visit exam.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, CRD Vision Care, Study Director — Alcon Research, LLC
Locations (8):
- United States (8):
  - Complete Family Vision Care, San Diego, California
  - Pearle Vision, Jacksonville, Florida
  - Jackson Health Community Center, Miami, Florida
  - Vision Health Institute, Orlando, Florida
  - Complete Eye Care of Medina, Medina, Minnesota
  - Koetting Associates, St Louis, Missouri
  - Sacco Eye Group, Vestal, New York
  - Smith Bowman Ophthalmology, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No